CLINICAL TRIAL: NCT03216551
Title: Evaluation of the Mediastinal Staging Accuracy of a Selective Lymphadenectomy Strategy Based on Tumor Location, Ground Glass Opacity Component and Frozen Section Diagnosis in Peripheral cT1N0M0 Invasive Non-small Cell Lung Cancer
Brief Title: Mediastinal Staging Accuracy of a Selective Lymphadenectomy Strategy in Early Stage NSCLC (ECTOP-1003)
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Professor, Fudan University
Other Study IDs: SASLND
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Lymph Node Metastases; Non-small Cell Lung Cancer Stage I
Keywords: selective mediastinal lymphadenectomy; minimally invasive surgery
MeSH Terms: conditions — Lymphatic Metastasis; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The assumed selective lymph node dissection group: Patients with consolidation tumor ratios ≤ 0.5 tumors will be considered to have negative mediastinal metastasis. Patients with intraoperative lepidic predominant adenocarcinoma diagnosis will be considered to have negative mediastinal metastasis. Patients with an apical tumor will be considered to have negative inferior mediastinal lymph node metastasis. If both N1 nodes and visceral pleural invasion are negative, patients with peripheral non-apical-segment upper lobe tumors will be considered to have negative inferior medistinal lymph node metastasis. If N1 nodes are negative, patients with left superior segment tumors will be considered to have negative 4L lymph node metasis, and patients with left basal segment tumors will be considered to have negative superior mediastinal lymph node metastasis.
  Interventions: Diagnostic Test: Intra-operative frozen section

INTERVENTIONS:
Diagnostic Test: Intra-operative frozen section — Tumor histologic subtypes (whether it is lepidic predominant adenocarcinoma), N1 nodes metastasis (lymph nodes adjacent to the tumor will be sent to frozen section) and visceral pleural invasion will be determined by the intra-operative frozen section.

SUMMARY:
This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-1003. Systemic mediastinal lymphadenectomy is deemed indispensable in lung cancer surgery for accurate staging and complete resection. However, extensive lymphadenectomy in patients without nodal metastasis may not improve survival and would increase operative duration and cause damage to mediastinal structures.Therefore the precise selection of patients without mediastinal nodal metastasis is the key to avoid unnecessary lymphadenectomy.The investigator's previous retrospective study shows tumor location, ground glass opacity component and histological subtypes are important predictors of negative nodal status in specific mediastinal regions. The current prospective observational study is to further verify the mediastinal staging accuracy of this selective lymphadenectomy strategy.

DETAILED DESCRIPTION:
Background:

Complete lung cancer lymphadenectomy in patients without nodal metastasis may not improve survival and would increase operative duration and cause damage to mediastinal structures.The investigator's previous retrospective study of 2749 invasive NSCLC patients showed none of the 151 tumors with consolidation tumor ratios ≤ 0.5 had N2 disease. Tumors with lepidic predominant adenocarcinoma (LPA) histology had zero mediastinal nodal involvement. Tumors in the apical segment of upper lobes had zero inferior mediastinal nodal (IMLN) involvement. Only seven out of 740 (0.9%) peripheral upper lobe tumors had IMLN metastasis. Interestingly, all these seven tumors showed visceral pleural invasion. Among patients with left lower lobe tumors, if hilar nodes were negative, station 4L lymph node metastasis was not found in superior and basal segment tumors, and station 5/6 lymph node involvement was always absent in basal segment tumors.

The current prospective, multi-center, observational study is to verify the staging accuracy of a selective mediastinal lymphadenectomy strategy based on tumor location, ground glass opacity component and intraoperative histological subtyping by frozen section in patients with peripheral clinical T1N0M0 invasive non-small cell lung cancer.

Objectives:

Primary: To determine the mediastinal staging accuracy of the selective mediastinal lymphadenectomy strategy.

Secondary:

1. To determine the diagnostic accuracy of intraoperative adenocarcinoma histologic subtyping, N1 nodes metastasis and visceral pleural invasion by frozen section.
2. To determine the mediastinal lymph node metastasis rate in peripheral clinical T1N0M0 lung cancer with different histologic subtypes.
3. To evaluate the pattern of mediastinal nodal involvement of tumors in different lung segments.
4. To determine the mediastinal nodal status of tumors with different radiological features (pure ground glass opacity, mixed ground glass opacity and solid nodules).

Outlines:

1. All recruited patients will undergo systematic mediastinal lymph node dissection (lung resection can be segmentectomy, lobectomy, bilobectomy or pneumonectomy). For tumors in the left lungs, removal of mediastinal nodal stations 4, 5,6,7 and 8 are required. For tumors in the right lungs, removal of mediastinal nodal stations 2,4,7 and 8 are required. For lower lobe tumors, station 9 should also be removed. Stations 10/11/12 should routinely be dissected.
2. Stations 10/11 are subclassified as follows: Station 10a (the anterior region of the pulmonary veins), Station 10s (between azygos vein and the right upper lobe bronchus), Station 10p (in the posterior region of the right main bronchus for right-side tumors or between left main pulmonary artery and left main bronchus for left-side tumors), Station 11s (between right upper lobe bronchus and the intermediate bronchus), and Station 11i (between right middle lobe bronchus and right lower lobe bronchus).
3. Intraoperative frozen section analysis should determine whether the tumor is lepidic predominant adenocarcinoma, whether there are N1 nodes involvement (lymph nodes adjacent to the tumor should be sent to intraoperative frozen section), and whether there is viceral pleural invasion. However, intraoperative frozen section results will not affect the surgical predure. Every patient will receive systematic lymph node dissection.
4. By the assumed selective lymph node dissection strategy, patients with consolidation tumor ratios ≤ 0.5 tumors will be considered to have negative mediastinal metastasis. Patients with intraoperative LPA diagnosis will be considered to have negative mediastinal metastasis. Patients with an apical tumor will be considered to have negative IMLN metastasis. If both N1 nodes and visceral pleural invasion are negative, patients with peripheral non-apical-segment upper lobe tumors will be considered to have negative IMLN metastasis. If N1 nodes are negative, patients with left superior segment tumors will be considered to have negative 4L lymph node metastasis, and patients with left basal segment tumors will be considered to have negative superior mediastinal lymph node metastasis. The virtual mediastinal staging results of this selective lymph node dissection strategy will then be compared with the final staging results by the complete lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent must be signed
* Peripheral clinical stage T1N0M0
* Invasive non-small cell lung cancer as determined preoperatively or intraoperatively, excluding AIS/MIA
* Can be completely resected
* If there are multiple nodules, except the predominant nodule, other nodules should be pure GGO

Exclusion Criteria:

* Previous malignancy or lung surgery
* Previous induction therapy for the disease
* Intolerable to the surgery
* Incomplete mediastinal lymph node dissection or lymph node sampling

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with peripheral clinical stage T1N0M0 who intended to be treated by radical surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1076 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Mediastinal staging accuracy of the assumed selective lymph node dissection strategy | 2-3 weeks after the surgery until the final pathology results are reported.
  To compare the mediastinal staging results by the assumed selective lymph node dissection strategy and the final staging results by systematic lymph node dissection.

SECONDARY OUTCOMES:
The accuracy of determining lepidic predominant adenocarcinoma, N1 nodes metastasis and viceral pleural invasion by frozen section | 2-3 weeks after the surgery until the final pathology results are reported.
  The concordance rate of intraoperative histologic subtypes, N1 node metastasis and visceral pleural invasion compared to the final pathology.
The nodal metastasis pattern of tumors in different lung segments. | 2-3 weeks after the surgery until the final pathology results are reported.
  The mediastinal nodal metastasis pattern of tumors in different lung segments.
The nodal status of tumors with various CT appearance | 2-3 weeks after the surgery until the final pathology results are reported.
  The nodal status of tumors with CT appearance of pure ground glass opacity, sub-solid and solid nodules.
The lymph node metastasis rate of different histologic subytpes. | 2-3 weeks after the surgery until the final pathology results are reported.
  The lymph node metastasis rate of different adenocarcinoma subytypes, squmous cell carcinoma, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, MD,PhD, Study Director — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided